CLINICAL TRIAL: NCT02846324
Title: A Phase II Randomized, Placebo-Controlled Study of GBT440 to Evaluate the Safety, Tolerability, Pharmacokinetics and Effect on Hypoxemia in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Study to Evaluate the Safety and Tolerability of GBT440 Administered to Subjects With IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GBT440-006
Record Dates: First submitted 2016-07-07; First posted 2016-07-27 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Idiopathic Pulmonary Fibrosis; Hypoxemia
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Hypoxia | interventions — voxelotor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- GBT440 600 mg Dose (Experimental): Parts A and B
  Interventions: Drug: GBT440
- GBT440 900 mg Dose (Experimental): Part A
  Interventions: Drug: GBT440
- GBT440 1500 mg Dose (Experimental): Part B
  Interventions: Drug: GBT440
- Placebo (Placebo Comparator): Parts A and B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GBT440 — Capsules which contain GBT440 drug substance in Swedish orange
  Arms: GBT440 1500 mg Dose; GBT440 600 mg Dose; GBT440 900 mg Dose
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial in which eligible IPF subjects will be randomized to receive GBT440 or Placebo orally daily.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of IPF.
* Oxygen desaturation with exercise.
* Completion of the baseline 6MWT
* Weight ≥ 50 kg
* Male or female of child bearing potential willing and able to use highly effective methods of contraception from study start to 3 months after the last dose of study drug.

Exclusion Criteria:

* FEV1/FVC < 70%.
* Subjects on supplemental oxygen therapy at rest.
* History of other interstitial lung diseases.
* Significant polycythemia.
* Female who is breast-feeding or pregnant.
* Known current malignancy or history of malignancy within the last 2 years prior to screening.
* Use of cytotoxic and/or immunosuppressant medications within 30 days screening.
* Hospitalization due to an exacerbation of IPF within 30 days of screening
* Subject plans to begin or has commenced pulmonary rehabilitation within 30 days of screening
* Corticosteroids (> 10 mg per day of prednisone or an equivalent) within 30 days of screening.
* Current smoker or history of smoking within 3 months of screening.
* Currently or, in the opinion of the investigator, soon to be listed for lung transplant.
* History of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within 6 months of screening.
* Any condition possibly affecting drug absorption.
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days or 5-half-lives, whichever is longer, prior to screening, or is currently participating in another trial of an investigational drug (or medical device).
* Subject who, for any reason, is deemed by the investigator to be inappropriate for this study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Birmingham, Alabama
  - San Francisco, California
  - Denver, Colorado
  - Miami, Florida
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - New York, New York
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Salt Lake City, Utah
  - Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GBT440 600 mg Dose | GBT440 900 mg Dose | GBT440 1500 mg Dose | Placebo
Started | 9 | 6 | 14 | 10
Completed Study Treatment | 7 | 5 | 11 | 10
Completed (Completed Study) | 7 | 6 | 10 | 10
Not Completed | 2 | 0 | 4 | 0
Not completed — Other | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- GBT440 600 mg Dose: Parts A and B Dose 1
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 900 mg Dose: Part A Dose 2
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 1500 mg Dose: Part B Dose 2; Overall Dose 3
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- Total: Total of all reporting groups
Arm/Group | Placebo | GBT440 600 mg Dose | GBT440 900 mg Dose | GBT440 1500 mg Dose | Total
Number analyzed (Participants) | 10 | 9 | 6 | 14 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (5.06) | 72.1 (6.31) | 65.7 (9.35) | 69.5 (5.67) | 69.8 (6.41)
Age, Continuous [Median (Full Range); unit: years] | 71.0 [62 to 77] | 72.0 [62 to 80] | 64.5 [56 to 77] | 69.5 [54 to 76] | 71.0 [54 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 3 | 8
  Male | 9 | 6 | 5 | 11 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 6 | 14 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 00 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 9 | 6 | 14 | 39
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.03
Time Frame: Days 1 to 58
Population: Participant had at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- GBT440 900mg Dose: Part A Dose 2
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 1500mg Dose: Part B Dose 2; Overall Dose 3
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
Arm/Group | Placebo | GBT440 600 mg Dose | GBT440 900mg Dose | GBT440 1500mg Dose
Number analyzed (Participants) | 10 | 9 | 6 | 14
Participants | 8 | 7 | 4 | 11

2. Secondary Outcome: Pharmacokinetic Profile of GBT440 Including Maximum Concentration
Time Frame: Days 1 and 28: pre-dose, and 2 hours post dose (+/- 15 minutes); Day 2: 24 hours (+/- 2 hours) after the Day 1 dose and prior to receiving the Day 2 dose; Days 8 & 15: pre-dose only
Population: Complete PK data was not analyzable for any participant.
Arm/Group | Placebo | GBT440 600 mg Dose | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic Profile of GBT440 Including Minimum Concentration
Time Frame: as for outcome 2
Population: Per protocol, analysis was to be conducted on complete PK analysis population; insufficient number of samples collected for pre-specified analysis.
Arm/Group | Placebo | GBT440 600 mg Dose | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetic Profile of GBT440 Including Apparent Terminal Half Life
Time Frame: as for outcome 2
Population: Complete PK data were not analyzable for any participant.
Arm/Group | Placebo | GBT440 600 mg Dose | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Evaluate the Effect of GBT440 on Oxygen Saturation Using Pulse Oximetry at Rest
Description: Data reported is change from baseline in Oxygen Saturation at rest
Time Frame: Baseline to Day 28
Measure: Least Squares Mean (Standard Error); unit: percent oxygen (%)
Groups:
- GBT440 Dose 1: Parts A and B
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 Dose 2: Part A
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 Dose 3: Part B
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
Arm/Group | Placebo | GBT440 Dose 1 | GBT440 Dose 2 | GBT440 Dose 3
Number analyzed (Participants) | 10 | 9 | 6 | 12
percent oxygen (%) | -1.1 (0.59) | 0.3 (0.77) | 0.4 (0.76) | 0.9 (0.57)

6. Secondary Outcome: Evaluate the Effect of GBT440 on Oxygen Saturation Using Pulse Oximetry After Exercise
Description: Change from Baseline to Day 28 after 6MWT
Time Frame: Baseline to Day 28
Population: 6MWT
Measure: Least Squares Mean (Standard Error); unit: percent oxygen (%)
Groups:
- GBT440 Dose 1: Parts A and B Dose 1
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 Dose 2: Part A Dose 2
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 Dose 3: Part B Dose 2; Overall Dose 3
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
Arm/Group | Placebo | GBT440 Dose 1 | GBT440 Dose 2 | GBT440 Dose 3
Number analyzed (Participants) | 10 | 9 | 6 | 12
percent oxygen (%) | -1.7 (1.64) | 2.9 (2.11) | 3.5 (2.16) | 3.5 (1.56)

ADVERSE EVENTS:
Time Frame: Screening to Day 58
Arm/Group | Placebo | GBT440 600 mg Dose | GBT440 900 mg Dose | GBT440 1500 mg Dose
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/9 | 1/6 | 2/14
Other Adverse Events (participants affected / at risk) | 8/10 | 7/9 | 4/6 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | GBT440 600 mg Dose (N=9) | GBT440 900 mg Dose (N=6) | GBT440 1500 mg Dose (N=14)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 2
Chronic myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Rash maculo papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Grade 3
Arterial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 3
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | GBT440 600 mg Dose (N=9) | GBT440 900 mg Dose (N=6) | GBT440 1500 mg Dose (N=14)
bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 5
nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 4
abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
flatulent (Gastrointestinal disorders) | 0 | 0 | 0 | 2
vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1
abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
dental carries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
fatigue (General disorders) | 1 | 1 | 1 | 2
pyrexia (General disorders) | 0 | 0 | 1 | 2
chills (General disorders) | 0 | 0 | 0 | 1
malaise (General disorders) | 0 | 0 | 0 | 1
oedema peripheral (General disorders) | 0 | 0 | 1 | 0
oedema (General disorders) | 1 | 0 | 0 | 0
drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
immunosuppression (Immune system disorders) | 0 | 1 | 0 | 0
sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
viral infection (Infections and infestations) | 0 | 0 | 0 | 1
viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
alanine immunotransferase increase (Investigations) | 0 | 0 | 0 | 1
aspartate immunotransferase increase (Investigations) | 0 | 0 | 0 | 1
eosinophil count increase (Investigations) | 0 | 0 | 0 | 1
gamma/glutamyltransferase increase (Investigations) | 1 | 0 | 0 | 1
lymph node palpable (Investigations) | 0 | 0 | 0 | 1
oxygen saturation decrease (Investigations) | 1 | 0 | 1 | 0
platelet count increase (Investigations) | 0 | 0 | 1 | 0
urine leukocyte esterase (Investigations) | 0 | 1 | 0 | 0
weight decreased (Investigations) | 0 | 0 | 0 | 1
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
headache (Nervous system disorders) | 0 | 1 | 0 | 2
dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0
insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
bilirubinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02846324/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02846324/SAP_001.pdf